CLINICAL TRIAL: NCT01686438
Title: Telemedicine Management of Veterans With PTSD and Chronic Insomnia
Brief Title: Telemedicine Management of Chronic Insomnia
Acronym: VIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 11-296
Record Dates: First submitted 2012-09-06; First posted 2012-09-18 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-07

CONDITIONS: Sleep Initiation and Maintenance Disorders; Post-Traumatic Stress Disorders
Keywords: cost effectiveness; patient satisfaction
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic; Patient Satisfaction | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT-I delivery by video teleconferencing (Experimental): Groups of participants will receive a cognitive behavioral therapy for insomnia program delivered by a trained psychologist using video teleconferencing.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia
- In-person CBT-I delivery (Active Comparator): Groups of participants will receive a cognitive behavioral therapy for insomnia (CBT-I) program by meeting in-person with a trained psychologist.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia — A behavioral modification program consisting of 6 clinic sessions focused on sleep hygiene, stimulus control, sleep restriction, and cognitive restructuring.
  Other Names: CBT-I

SUMMARY:
Insomnia is commonly present in Veterans with post-traumatic stress disorder (PTSD). Treatment of insomnia with a specialized type of psychotherapy has been shown to be more effective than treatment with medications. Unfortunately, few psychologists are trained to provide this treatment, limiting Veterans' access to care, especially those Veterans in remote and rural areas. This project will evaluate the ability to deliver this psychotherapy to groups of Veterans by video teleconferencing. Groups of Veterans with PTSD and chronic insomnia will receive the psychotherapy treatment either by meeting in-person with the psychologist or by the psychologist delivering the treatment by video teleconferencing. Finding that video teleconferencing is a cost effective way to deliver this treatment could add an important new component to the care of Veterans with PTSD that provides an alternative to medications.

DETAILED DESCRIPTION:
Objectives(s): The investigators are conducting a randomized, controlled trial of Veterans with PTSD and chronic insomnia to determine if cognitive behavioral therapy for insomnia (CBT-I) administered by video teleconferencing is not clinically inferior to in-person treatment in terms of improvement in insomnia symptoms. Secondary aims are 1) comparing the differences in cost and quality-adjusted life years between the treatment delivery approaches and 2) determining the effectiveness of CBT-I on functional outcomes, sleep quality, and non-sleep-related PTSD symptoms. The investigators are also conducting a patient- and provider-focused formative evaluation of CBT-I delivery by video teleconferencing to assess potential barriers to its widespread implementation.

Research Design: This prospective randomized controlled non-inferiority study will determine if Veterans with PTSD and chronic insomnia receiving CBT-I by video teleconferencing have an improvement in insomnia severity, as determined by change in Insomnia Severity Index (ISI) score, that is not clinically inferior to that in Veterans receiving in-person CBT-I. Differences in cost and quality-adjusted life years (QALY) between groups will also be compared.

Methodology: Veterans with PTSD and chronic insomnia receiving their primary care at community-based outpatient clinics (CBOC) affiliated with the Philadelphia VAMC are be randomized to receive one of the following interventions in a group setting at their CBOC: 1) a manual-based CBT-I program delivered via video teleconferencing, 2) the CBT-I program delivered in-person, and 3) in-person delivery of sleep hygiene education, a known active control intervention. Participants are assessed at baseline, and 2 weeks and every 3 months following the intervention. The primary outcome measure in Aim 1 is the change in the Insomnia Severity Index (ISI) score at 6 months following intervention. Non-inferiority analysis will be used to compare the effectiveness of the two delivery methods, with a pre-specified margin. Results will be ascertained via intent to treat and per-protocol procedures. The investigators hypothesize that the change in ISI score following CBT-I by video teleconferencing will not be clinically inferior to that following in-person delivery. In Aim 2, VA and non-VA total healthcare costs are being collected to test whether average cost is lower for Veterans receiving CBT-I by video teleconferencing versus in-person care. Preference is being assessed by the EuroQol and Health Utilities Index 2. Differences in the ratio of cost and quality-adjusted life years saved between CBT-I by video teleconferencing and in-person encounter will be compared to test the hypothesis that video teleconferencing will have lower cost and equivalent outcomes. Aim 3 is assessing the effect of CBT-I on functional outcomes (Short Form-12, Work and Social Adjustment Scale), sleep quality (Pittsburgh Sleep Quality Index, sleep diary and wrist actigraphy), and PTSD severity (the non-sleep component of the PTSD Checklist-Military). The investigators hypothesize that these functional outcomes and sleep quality measures will improve following each method of CBT-I delivery and that CBT-I will improve non-sleep-related PTSD severity. The formative evaluation of the telemedicine delivery of CBT-I in Aim 4 is using qualitative (targeted focus groups with participants and therapist interviews) and quantitative measures (Work Alliance Inventory, Treatment Credibility Scale, attrition) that will help guide future implementation of CBT-I by video teleconferencing

Anticipated Findings: The investigators believe these results will demonstrate that: 1) Veterans in both CBT-I groups will have similar improvement in functional outcomes, and 2) treatment delivery by video teleconferencing will be more cost effective than in-person care. These findings should lead to wider acceptance of video teleconferencing, thereby increasing patient access to care and reducing treatment costs.

ELIGIBILITY:
Inclusion Criteria:

Veterans will have to meet the following inclusion criteria in order to be enrolled in this RCT:

* Men and women at least 18 years of age.
* Meet current DSM-IV-TR criteria for PTSD as determined by the Clinician Administered PTSD Scale (CAPS)
* Insomnia Severity Index score > 14, the commonly used threshold for clinical insomnia, with self-reported duration of insomnia >6 months.
* Ability to read and speak English (assessment instruments and therapy will be available only in English)

Exclusion Criteria:

Veterans will be excluded from participation if they meet any of the following exclusion criteria:

* Unable or unwilling to provide informed consent.
* Unwilling to participate in supervised group sessions at the community based outpatient clinic
* No telephone access or inability to return for follow-up testing.
* Individuals with an untreated sleep disorder [e.g., obstructive sleep apnea (apnea-hypopnea index 15 events/hr), periodic limb movement disorder (10 leg movements/hr of sleep with arousals), central sleep apnea ( 50% of apneas are central), Cheyne-Stokes respiration, obesity hypoventilation syndrome, and narcolepsy].
* A clinically unstable medical condition as defined by a new diagnosis or change in medical management in the previous 2 months.
* Evidence of substance dependence during the preceding twelve months. Evidence of "at risk" drinking behavior over the past month. Namely for men: more than 4 drinks on a given night, drinking on more than 3 nights a week, or more than 14 total drinks in a week; for women: more than 3 drinks in a given night, drinking on more than 3 nights a week, or more than 7 total drinks in a week.
* Individuals with bipolar disorder, delirium, dementia, amnestic disorder, schizophrenia and other psychotic disorders as determined by the SCID questionnaire. A concurrent anxiety disorder or depressive disorder diagnosis will be allowed.
* Individuals with prominent current suicidal or homicidal ideation. This will be assessed by the clinical psychologist administering the SCID and CAPS. In cases of prominent current suicidal or homicidal ideation appropriate safety measures will be taken. Following stabilization, Veterans who continue to be interested in participating in the study may be re-assessed.
* Unable to perform tests due to inability to communicate verbally, inability to read and write; less than a 5th grade reading level; visual, hearing or cognitive impairment (e.g., previous head injury).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T. Kuna, MD, Principal Investigator — Philadelphia VA Medical Center, Philadelphia, PA
Locations (1):
- Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gehrman P, Shah MT, Miles A, Kuna S, Godleski L. Feasibility of Group Cognitive-Behavioral Treatment of Insomnia Delivered by Clinical Video Telehealth. Telemed J E Health. 2016 Dec;22(12):1041-1046. doi: 10.1089/tmj.2016.0032. Epub 2016 Jun 10. PMID 27286369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 114 participants were consented and randomized in the study. 87 of those participants started in treatment in this study. Of those, 57 completed treatment sessions. 55 of the 57 who completed treatment are included in the analysis of this study.
Groups:
- Control: Non-active intervention of sleep education delivered in-person
- CBT-I In-person: Cognitive behavior therapy for insomnia (CBT-I) delivered in-person
- CBT-I Telehealth: Cognitive behavior therapy for insomnia (CBT-I) delivered via video teleconferencing
Period: Overall Study
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Started | 15 | 35 | 37
2-Week Follow Up | 12 | 31 | 27
3-Month Follow Up | 7 | 21 | 17
6-Month Follow Up | 7 | 26 | 24
Completed | 7 | 26 | 24
Not Completed | 8 | 9 | 13
Not completed — Lost to Follow-up | 8 | 9 | 10
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: patients who attended over 3 sessions and had a non-missing 3 month visit
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth | Total
Number analyzed (Participants) | 7 | 25 | 23 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.57 (10.05) | 56.16 (10.84) | 56.57 (11.24) | 56.89 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 0 | 6
  Male | 6 | 20 | 23 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4 | 12 | 11 | 27
  Black or African American | 3 | 11 | 9 | 23
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Unavailable (do not wish to provide information) | 0 | 2 | 2 | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.05 (2.79) | 34.02 (6.77) | 34.31 (4.97) | 33.89 (5.64)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Insomnia Severity Index Score
Description: Self-report questionnaire used widely to assess presence of insomnia and its severity. Scores range from 0-28. Higher scores indicate increasing severity of insomnia.
Time Frame: Baseline to 3 months
Population: Participants who attended over 3 sessions and had a non-missing 3 month visit (all available observations). This analysis was intended to only compare the two CBT-I groups for non-inferiority analysis.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 25 | 23
units on a scale | 6.68 (1.09) | 5.13 (1.15)
Statistical Analysis 1: Comparison: CBT-I In-person vs CBT-I Telehealth; Test type: Non-Inferiority — The mean change in ISI score from baseline in Veterans receiving CBT-I by video teleconferencing will be no more than 1.67 smaller than the reference treatment, i.e., Veterans receiving in-person CBT-I; p = 0.138, t-test, 1 sided; Mean Difference (Net) = -2.03, 95% CI 2-sided [-4.63 to 1.57], Standard Deviation 1.33

2. Secondary Outcome: Change From Baseline PTSD Checklist-Military (PCL-M) Scores
Description: Self-administered validated questionnaire measuring PTSD severity. Scores range from 17-85. Higher scores indicate higher severity of symptoms.
Time Frame: baseline to 3 months
Population: Participants who attended over 3 sessions and had a non-missing 3 month visit (all available observations
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
units on a scale | 3.30 (3.33) | 5.73 (1.87) | 5.22 (1.96)

3. Secondary Outcome: Change From Baseline Pittsburgh Sleep Quality Index (PSQI) Scores
Description: Self-administered validated questionnaire measuring subjective sleep quality. Scores range from 0-21. Higher score indicates worse sleep quality. Total score < 5 is associated with good sleep quality.
Time Frame: baseline to 3 months
Population: Participants who attended over 3 sessions and had a non-missing 3 month visit (all available observations)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
units on a scale | 2.03 (1.36) | 3.34 (0.71) | 2.50 (0.76)

4. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index Addendum for PTSD (PSQI-A)
Description: Measure of the sleep and dream disturbances often associated with PTSD. Scores range from 0-21. A higher score indicates higher frequency of disruptive nocturnal behaviors. Total score ≥ 4 can be used to indicate PTSD.
Time Frame: baseline to 3 months
Population: Patients who attended over 3 sessions and had a non-missing 3 month visit (all available observations)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
units on a scale | 0.30 (1.13) | 0.23 (0.66) | 0.51 (0.71)

5. Secondary Outcome: Change From Baseline in Nightmare Distress Questionnaire Scores
Description: Measure of intensity of the distress associated with a nightmare. Scores range from 0-52. Higher score indicates increased nightmare distress.
Time Frame: baseline to 3 month
Population: Participants who attended over 3 sessions and had a non-missing 3 month visit (all available observations)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
units on a scale | -3.78 (1.67) | -2.65 (0.98) | -0.11 (1.07)

6. Secondary Outcome: Change From Baseline Medical Outcomes Study Short Form-12 (SF-12) Mental Component Score
Description: Self-administered validated general health-related quality of life questionnaire to assess functional outcome. Scores range from 0 to 100. Higher scores indicate higher health function.
Time Frame: baseline to 3 months
Population: Participants who attended over 3 sessions and had a non-missing 3 month visit (all available observations)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
units on a scale | 0.26 (2.79) | 0.70 (1.55) | 2.76 (1.65)

7. Secondary Outcome: Change From Baseline in Medical Outcomes Study Short Form-12 (SF-12) Physical Component Score
Description: self-administered validated health related quality of life questionnaire to assess functional outcomes. Scores range from 0 to 100. Higher scores indicate higher health function.
Time Frame: baseline to 3 months
Population: patients who attended over 3 sessions and had a non-missing 3 month visit (all available observations)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
units on a scale | 3.31 (2.24) | -1.37 (1.22) | 0.14 (1.31)

8. Secondary Outcome: Change From Baseline in Work and Social Adjustment Scale Scores
Description: A self-report scale of functional impairment attributable to an identified problem. Scores range from 0 - 40. Higher scores indicate increasing functional impairment.
Time Frame: baseline to 3 months
Population: Participants who attended over 3 sessions and had a non-missing 3 month visit (all available observations)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
units on a scale | -0.54 (2.77) | 0.01 (1.46) | -0.85 (1.63)

9. Secondary Outcome: Working Alliance Inventory - Short Revised (WAI-SR) - Task Formation Scores at 8 Weeks
Description: The WAI-SR is a 12 item self report of patient's perceived quality of interaction with practitioner. The scale focuses on task alliance, goal alliance, and bond formation. Items range from 1- never to 7- always. Scores range from 7-84. Higher scores indicate better alliance. Scores are reported from session 4.
Time Frame: 2-8 weeks
Population: patients who attended over 3 sessions and had a non-missing 3 month visit (all available observations)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
score on a scale | 62.5 (6.24) | 76.8 (5.02) | 74.1 (8.64)

10. Secondary Outcome: Charleston Psychiatric Outpatient Satisfaction Scale-VA Scores at 8 Weeks
Description: Self administered questionnaire of person's satisfaction with care. Total scores range from 13 to 65, with higher scores indicating higher patient satisfaction. Scores reported from session 5.
Time Frame: 2-8 weeks
Population: patients who attended over 3 sessions and had a non-missing 3 month visit (all available observations)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
score on a scale | 47.5 (6.54) | 46.7 (9.09) | 44.8 (12.16)

11. Secondary Outcome: Change From Baseline in Nightmare Frequency Questionnaire (NFQ) Part 1 Scores
Description: Measure of nightmare frequency in number of nights with nightmares per year, scores converted to yearly.
Time Frame: baseline to 3 months, scores converted to yearly
Population: Participants who attended over 3 sessions and had a non-missing 3 month visit (all available observations), converted scores to yearly.
Measure: Least Squares Mean (Standard Error); unit: nights per year
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
nights per year | -26.1 (20.13) | 11.35 (11.39) | -3.04 (12.65)

12. Secondary Outcome: Change From Baseline in Nightmare Frequency Questionnaire (NFQ) Part 2 Scores
Description: Self-administered measure of nightmare frequency in actual number of nightmares experienced over a 3 month period, and converted to yearly
Time Frame: baseline to 3 months (converted to yearly)
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: number of nightmares
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
number of nightmares | -24.6 (23.87) | 6.41 (13.48) | -8.09 (15.27)

13. Secondary Outcome: Working Alliance Inventory - Short Revised (WAI-SR) - Bond Formation at 8 Weeks
Description: as for outcome 9
Time Frame: 2-8 weeks
Population: patients who attended over 3 sessions and had a non-missing 3 month visit (all available observations)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
score on a scale | 72.8 (11.15) | 77.4 (7.57) | 76.8 (8.41)

14. Secondary Outcome: Working Alliance Inventory - Short Revised (WAI-SR) - Goal Formation at 8 Weeks
Description: as for outcome 9
Time Frame: 2-8 weeks
Population: patients who attended over 3 sessions and had a non-missing 3 month visit (all available observations)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Number analyzed (Participants) | 7 | 25 | 23
score on a scale | 67.5 (10.15) | 75.8 (7.54) | 75.3 (10.28)

ADVERSE EVENTS:
Time Frame: Duration of study, an average of 2.5 years
Arm/Group | Control | CBT-I In-person | CBT-I Telehealth
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/35 | 1/37
Other Adverse Events (participants affected / at risk) | 0/15 | 2/35 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=15) | CBT-I In-person (N=35) | CBT-I Telehealth (N=37)
hospitalized for suicide ideation (Psychiatric disorders) | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=15) | CBT-I In-person (N=35) | CBT-I Telehealth (N=37)
Tonsillectomy (Surgical and medical procedures) | 0 | 1 (1) | 0
Gout (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes